CLINICAL TRIAL: NCT02571348
Title: Optimum Micro-osteoperforations Accelerated Tooth Movement Interval, Related Pain Perception and Impact to Daily Functions - A Randomized Controlled Trial
Brief Title: Optimum Micro-osteoperforations Accelerated Tooth Movement Interval
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DF CD1412/0089(P)
Record Dates: First submitted 2015-10-05; First posted 2015-10-08 (Estimated); Last update posted 2016-12-30 (Estimated); Status verified 2016-12

CONDITIONS: Accelerated Tooth Movement Interval

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 4 weeks and 8 weeks (Active Comparator): Micro-osteoperforation will be done on either side of the maxilla at 4 weeks interval and the contralateral site will be the control. In mandible, micro-osteoperforation will be done every 8 weeks and the contralateral site will serve as the control
  Interventions: Procedure: micro-osteoperforation
- 8 weeks and 12 weeks (Active Comparator): Micro-osteoperforation will be done on either side of the maxilla at 8 weeks interval and the contralateral site will be the control. In mandible, micro-osteoperforation will be done every 12 weeks and the contralateral site will serve as the control
  Interventions: Procedure: micro-osteoperforation
- 12 weeks and 4 weeks (Active Comparator): Micro-osteoperforation will be done on either side of the maxilla at 12 weeks interval and the contralateral site will be the control. In mandible, micro-osteoperforation will be done every 4 weeks and the contralateral site will serve as the control
  Interventions: Procedure: micro-osteoperforation

INTERVENTIONS:
Procedure: micro-osteoperforation — micro-osteoperforation with mini implant at different interval

SUMMARY:
This study is intended to investigate the optimum interval between micro-osteoperforations to accelerate orthodontic tooth movement. Overall, the investigator will be comparing the rate of tooth movement between micro-osteoperforated site and non micro-osteoperforated site. Next, the investigator will be comparing the rate of orthodontic tooth movement for micro-osteperforation performed at 4, 8 and 12 weeks' intervals. In addition, the investigator will be evaluating the pain intensity and impact of pain on quality of life during different intervals of micro-osteoperforations at 4, 8 and 12 weeks. Finally, the investigator will be comparing the rate of orthodontic tooth movement between maxilla and mandible.

The significance of the outcome is to determine optimum recommended interval for micro-osteopeforation which can be used to accelerate orthodontic tooth movement. By finding out the optimum interval, the investigator can come with a recommended interval of micro-osteoperforation which can be used routinely in patients to fasten orthodontic tooth movement.

DETAILED DESCRIPTION:
1. TRIAL DESIGN This is a prospective randomized clinical trial and single centre study (Faculty of Dentistry, University of Malaya). Participants included are molar class I malocclusion, molar Class II & III < ½ unit, requiring extraction of all four permanent first premolar and maximum anchorage control with Temporary Anchorage Device (TAD).
2. SAMPLE SIZE CALCULATION Sample size calculation is based on a type 1 error frequency of 5% and the power of the statistical test set at 90% ( P = 0.9, B = 0.1 ) This is based on animal study as a guide to detect at least 50% difference in the rate of tooth movement. ( Teixeira CC et al.,2010). The sample size was calculated based on a formula described by Lisa Kuramoto from Vancouver Coastal Health Research Institute. Total participant needed with be 30 with minimum of 10 participants per group. We anticipate 20% drop-outs based on previous study. Thus, a minimum of 36 participants will be recruited.

4. ETHICAL APPROVAL Approval for the conduct of this study had been obtained from Medical Ethics Committee, University of Malaya 5. RANDOMIZATION This study will be conducted by one orthodontic resident together with one orthodontic Consultant from Faculty of Dentistry, University Malaya, who is the main supervisor of this study. A simple randomization method will be employed to assign patient into experimental site and also the for the frequency interval of micro-osteoperforation.

6. INTERVENTION Sequence of events during clinical trial is as follows:-

1. Diagnostic record taking (Study models, Photographs, and x-ray)
2. Randomization for experimental sites in maxilla and mandible & randomization for interval of micro-osteoperforation (Group 1: 4weeks maxilla & 8weeks mandible, Group 2: 8weeks maxilla & 12weeks mandible, Group 3: 12 weeks maxilla & 4 weeks mandible)
3. Treatment planning with Orthodontic Consultant
4. Placement of TADs bilaterally in maxilla and mandible & Clinical calibration for inter-observer error
5. Referral for extraction of 14,24,34 and 44 (Extraction must be done within 2 weeks after insertion of TADs)
6. One month after extraction, Banding and Bonding of upper and lower preadjusted edgewise fixed appliances (MBT prescription 0.022"x 0.028" slot).
7. Arch wire sequence for levelling and aligning are as follows:-

   * Upper and lower 0.014 NiTi Arch wire
   * Upper and lower 0.018 NiTi Arch wire
   * Upper and lower 17 x 25 NiTi Arch wire
   * Upper and lower 19 x 25 SS Arch wire

     * Dead coil will be placed to maintain the extraction space of premolars
     * Interval between each arch wire sequence is 6 weeks
8. One month after the insertion of working arch wire, micro-osteoperforations will be performed & Inter-obverver error measurement will be done 2 weeks after insertion of working arch wire and on the day of mirco-osteoperforations.
9. Three micro-osteoperforations will be placed at the buccal aspect on the buccal cortical bone at the site of premolar extraction(experimental site only) and both canine will be retracted bilaterally with NiTi Coil Spring.
10. Participants will be given questionnaire after the procedure and the questionnaire will be collected the following visit 11 From now onwards, participants will be reviewed at their respective interval. Either 4,8 or 12 weeks interval.

12. This is the critical period of this study in which micro-osteoperforations will be performed and questionnaire will be given to participants.

13. Data collection will be conducted for a period of 16weeks(4 months) - during canine retraction

ELIGIBILITY:
Inclusion Criteria:

* Molar Class I malocclusion, molar Class II & III < ½ unit, requiring extraction of all four permanent first premolar and maximum anchorage control with temporary anchorage device (TAD)
* Average vertical facial proportions
* No systemic disease
* Good oral hygiene
* No history of periodontal therapy
* No current active periodontal disease

Exclusion Criteria:

* Vertical skeletal discrepancies eg high angle and low angle
* Systemic disease especially on long term use of antibiotics, phenytoin, cyclosporin, anti-inflammatory drugs, systemic corticosteroid and calcium channel blockers
* Poor oral hygiene for more than 3 visits
* Past periodontal disease
* Current periodontal disease

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
rate of orthodontic tooth movement between micro osteoperforated site and non micro-osteoperforated site. | through study completion, an average of 2 years

SECONDARY OUTCOMES:
Rate of orthodontic tooth movement between maxilla and mandible. | through study completion, an average of 2 years
Rate of orthodontic tooth movement when micro-osteperforation performed at 4, 8 and 12 weeks intervals. | through study completion, an average of 2 years
Pain intensity and impact of pain on patient's daily functions during different intervals of micro-osteoperforations at 4, 8 and 12 weeks using questionnaire. | through study completion, an average of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Wey Mang Check, Principal Investigator — Faculty of Dentistry, University of Malaya; Jennifer Geraldine Doss, Principal Investigator — Faculty of Dentistry, University of Malaya; Saritha Sivarajan, Principal Investigator — Faculty of Dentistry, University of Malaya
Locations (1):
- Faculty of Dentistry, University of Malaya, Kuala Lumpur, Kuala Lumpur, Malaysia

REFERENCES:
- [Result] Alikhani M, Khoo E, Alyami B, Raptis M, Salgueiro JM, Oliveira SM, Boskey A, Teixeira CC. Osteogenic effect of high-frequency acceleration on alveolar bone. J Dent Res. 2012 Apr;91(4):413-9. doi: 10.1177/0022034512438590. Epub 2012 Feb 14. PMID 22337699
- [Result] Teixeira CC, Khoo E, Tran J, Chartres I, Liu Y, Thant LM, Khabensky I, Gart LP, Cisneros G, Alikhani M. Cytokine expression and accelerated tooth movement. J Dent Res. 2010 Oct;89(10):1135-41. doi: 10.1177/0022034510373764. Epub 2010 Jul 16. PMID 20639508
- [Result] Krishnan V, Davidovitch Z. On a path to unfolding the biological mechanisms of orthodontic tooth movement. J Dent Res. 2009 Jul;88(7):597-608. doi: 10.1177/0022034509338914. PMID 19641146
- [Result] Krishnan V, Davidovitch Z. Cellular, molecular, and tissue-level reactions to orthodontic force. Am J Orthod Dentofacial Orthop. 2006 Apr;129(4):469.e1-32. doi: 10.1016/j.ajodo.2005.10.007. PMID 16627171
- [Result] Ren Y, Kuijpers-Jagtman AM, Maltha JC. Immunohistochemical evaluation of osteoclast recruitment during experimental tooth movement in young and adult rats. Arch Oral Biol. 2005 Dec;50(12):1032-9. doi: 10.1016/j.archoralbio.2005.04.005. Epub 2005 Jun 15. PMID 15963453
- [Result] Long H, Pyakurel U, Wang Y, Liao L, Zhou Y, Lai W. Interventions for accelerating orthodontic tooth movement: a systematic review. Angle Orthod. 2013 Jan;83(1):164-71. doi: 10.2319/031512-224.1. Epub 2012 Jun 21. PMID 22720793